CLINICAL TRIAL: NCT01007058
Title: Markers of Response to Intravesical Bladder Cancer Therapy
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Flight Attendant Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LAB05-0326
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Bladder Cancer
Keywords: Urinary Bladder; Non-muscle-invasive transitional cell carcinoma; Intact bladder; Intravesical Bladder Cancer Therapy; Tumor Recurrence; Surrogate markers of response; BCG; Bacillus Calmette Guérin; Interferon-alfa-2b; IFN-alfa-2b; Interferon; Fluorescence in situ hybridization; FISH
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4 tablespoons of urine and a bladder wash sample during catheterization (for planned treatment) or during routine cystoscopic exam, both samples at 4 different time points before, during and after therapy courses.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Response Markers: Urine Collection and Bladder wash of Bladder Cancer Patients with Treatment of BCG or BCG plus interferon

SUMMARY:
The goal of this laboratory research study is to see if researchers can predict whose cancer will stay in remission and whose will return in patients receiving treatment for bladder cancer.

DETAILED DESCRIPTION:
In this study, researchers are looking at markers that they could use to identify - at an early time point - those patients who might not respond to this treatment. This would allow researchers to provide future patients with information about their chances of responding to such treatment. And, with this information, researchers could better counsel those patients who might benefit from a different therapy at an earlier time point.

Treatment with BCG or BCG plus interferon is currently the most effective nonsurgical treatment for superficial bladder cancer. However, at this time, there is no reliable test that can help researchers predict which patients will respond to this therapy. You will be receiving BCG or BCG plus interferon therapy as planned by your physician. This is a standard therapy that will be decided by your doctor and based on your disease characteristics. If you agree to take part in this study, your participation will not affect the treatment you will receive in any way. Your follow-up and disease monitoring will be done according to standard routines.

By participating in this study, you agree to provide researchers with 4 tablespoons (or as much as you can produce) of urine at the following time points.

1. Before you start therapy.
2. Just before and 4 hours after your last treatment (which usually occurs 6 weeks after start of treatment).
3. Just before and 4 hours after your last treatment of the second course of therapy (which is usually about 3 months after the beginning of the first course of therapy.

In addition, you will provide researchers with a bladder wash sample. This sample will be collected during routine catheterization (for your planned treatment) or during your routine cystoscopic exam. Bladder wash samples will be collected at the following time points.

1. Before you start therapy.
2. Just before your last treatment (which usually occurs 6 weeks after start of treatment).
3. At your first routine cystoscopic follow-up (which usually occurs at 3 months).
4. At your second routine cystoscopic follow-up (which usually occurs at 6 months).

Your follow-up cystoscopies and maintenance therapy will be done according to routine care as decided by your doctor and are not affected by your participation in this study. You will be part of the study for about 24 months after beginning the treatments. At the end of that period, between 23 and 27 months, you will be checked with cystoscopy and cytology to see if the tumor has come back, as part of standard of care.

In addition, information will be collected from your medical chart about other medications that you are taking and other conditions, such as diabetes or heart disease, that you may have. Information will also be collected about previous treatment that you have had for bladder cancer as well as other treatments that you may receive during this study. This may include treatments that are received at an outside health facility. Neither your name nor your medical record number will be kept with this information. All of the information collected for this study will be kept in a locked cabinet to which only the researchers have access. Upon completion of the study, the information sheets will be destroyed.

This is an investigational study.

A total of 300 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics:

* Histologically confirmed primary or recurrent non-muscle-invasive transitional cell carcinoma with an intact bladder
* Stage Ta, T1, or carcinoma in situ
* Grade 1, 2, or 3
* Primary disease site must be the urinary bladder
* No evidence of tumor invasion of the muscularis propria by cystoscopy and biopsy within the past 6 weeks
* Upper tract imaging within the prior 12 months

Patient Characteristics:

* Age: 18 years and above
* Gender: Male or female
* Life expectancy: 24 months or greater
* Performance status: 0 - 1

Prior Therapy:

* Biologic therapy: allowed
* Chemotherapy: allowed
* Radiotherapy: no prior pelvic radiotherapy
* Surgery: recovered from prior transurethral resection

Intravesical Immunotherapy:

* In the opinion of the treating physician, the patient must be a candidate for "standard of care" intravesical immunotherapy, defined as

  * Induction with 6 weekly treatments of intravesical BCG followed by maintenance with 3 weekly treatments of intravesical BCG at 3 months. Continued maintenance therapy at 6 months and then every 6 months for total of 36 months ("Lamm regimen") (38) is optional and left to the discretion of the physician or
  * Induction with 6 weekly treatments of intravesical BCG plus IFN-alfa-2b followed by maintenance with 3 weekly treatments of BCG plus IFN-alfa-2b at 3 months. Continued maintenance therapy at 9 months, and 15 months ("O'Donnell regimen") (39) is optional and left to the discretion of the physician.
* Patients will be included in the study based on 'intent to treat'. If, after start of induction, the treating physician decides to alter the treatment regimen, patients will still be included for analysis.

Special Situations:

A special situation arises when during the course of the study, a patient develops recurrent tumor, and is deemed by the treating physician to require either a reinduction course of BCG therapy or therapy with BCG plus Interferon. In that case, the patient will remain in the protocol and, since urine cytology/FISH and cytokine responses are dependent on the treatment time-table, we will start collecting urine samples all over again, as already described previously in the protocol. Also, starting from the change in the treatment plan, the patient's overall time in the protocol will be prolonged up to the completion of a 24-month period of time.

Exclusion Criteria

* Ongoing Pregnancy
* Patients who are not eligible to receive standard-of-care intravesical immunotherapy such as

  * histologically confirmed pure squamous cell carcinoma or pure adenocarcinoma,
  * patients with nonurothelial bladder cancer such as sarcoma, and immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients, 18 years or older, who will be receiving treatment with BCG or BCG + Interferon at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2005-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Clinical tumor recurrence or progression by 24 months after initiation of intravesical immunotherapy | Baseline to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ashish M. Kamat, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Kamat AM, Briggman J, Urbauer DL, Svatek R, Nogueras Gonzalez GM, Anderson R, Grossman HB, Prat F, Dinney CP. Cytokine Panel for Response to Intravesical Therapy (CyPRIT): Nomogram of Changes in Urinary Cytokine Levels Predicts Patient Response to Bacillus Calmette-Guerin. Eur Urol. 2016 Feb;69(2):197-200. doi: 10.1016/j.eururo.2015.06.023. Epub 2015 Jun 25. PMID 26119560
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org